CLINICAL TRIAL: NCT02133027
Title: Role of the Right Portal Pedicle and Rouviere's Sulcus as an Anatomic Landmark in Laparoscopic Cholecystectomy in Chinese Population
Brief Title: Role of the Right Portal Pedicle and Rouviere's Sulcus as an Anatomic Landmark in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fanyingfang3
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Gallstones; Cholecystitis; Polyps
Keywords: Laparoscopic cholecystectomy
MeSH Terms: conditions — Gallstones; Cholecystitis; Polyps | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rouviere's Sulcus (Experimental): Rouviere's sulcus is a 2 to 5 cm sulcus running to the right of the liver hilum anterior to the caudate process and usually containing the right portal triad or its branches.Dissection may be started safely by division of the peritoneum immediately ventral to the sulcus and continued in a triangle bounded by the liver surface, the neck of the gallbladder and the plane of the sulcus.
  Interventions: Procedure: Rouviere's sulcus; Device: surgical instruments
- traditional anatomy method (Other): Ratcheted grasper is inserted through the lateral 5-mm port to retract the gallbladder fundus in cephalad fashion. An atraumatic grasper is inserted through the middle 5-mm port to retract the gallbladder infundibulum laterally, exposing the anteromedial aspect of the triangle of Calot.
  Interventions: Device: surgical instruments

INTERVENTIONS:
Procedure: Rouviere's sulcus — Dissection may be started safely by division of the peritoneum immediately ventral to the sulcus and continued in a triangle bounded by the liver surface, the neck of the gallbladder and the plane of the sulcus.
  Arms: Rouviere's Sulcus
Device: surgical instruments — surgical instruments used in the laparoscopic cholecystectomy,such as ratcheted grasper,atraumatic grasper ,scissors.
  Other Names: Operating apparatus

SUMMARY:
Objective:To explore the role of the right portal pedicle and Rouviere's sulcus as an anatomic landmark in laparoscopic cholecystectomy.

Methods:The investigators are going to select 60 patients intending to perform Laparoscopic cholecystectomy from April 2014 to April 2015.Check out the presence of the right portal pedicle and Rouviere's sulcus during the surgery and divide into the experimental group and the control group.Experimental group operated in Laparoscopic cholecystectomy with the guide of Rouviere's sulcus while the Control group operated with the traditional way.

Research hypothesis:Compare the differences between the Experimental group and the Control group in bile duct injury rate,complication rate,blood loss,operative time ,conversion rate and hospital stay.It is supposed that the results of Experimental group are superior to the control group,difference is statistically significant(P<0.05). So the investigators can draw the conclusion that the anatomy method with the guide of right portal pedicle and Rouviere's sulcus is useful in laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Surgical procedures(Experimental group ):Placing the grasping forceps on the neck of the gallbladder, then retracted upwards and towards the left, so that the posterior aspect of the hepatobiliary triangle is exposed. the sulcus is seen running to the right of the hilum . In some patients, the lips of the sulcus are partially fused, with only a small cleft visible laterally. The sulcus indicates reliably the plane of the common bile duct; dissection may be started safely by division of the peritoneum immediately ventral to the sulcus and continued in a triangle bounded by the liver surface, the neck of the gallbladder and the plane of the sulcus. Even if the bile duct is tented upwards by the traction that has been exerted on the gallbladder, dissection will be safely ventral to the plane of the duct. Posterior branches of the cystic artery, may lie in the area of dissection and must be identified with care.Once a plane has been opened posteriorly, attention may be turned to the anterior dissection, using the posterior landmarks as a guide. The anterior and posterior dissections can then be made to meet, thus opening the hepatobiliary triangle completely.

Surgical procedures(Control group ):A small periumbilical incision is made, with the location and orientation depending on the patient's body habitus and cosmetic considerations.The laparoscope is used to explore the abdomen for adhesions and potential injuries that may have occurred during port placement，ratcheted grasper is inserted through the lateral 5-mm port to retract the gallbladder fundus in cephalad fashion. An atraumatic grasper is inserted through the middle 5-mm port to retract the gallbladder infundibulum laterally, exposing the anteromedial aspect of the triangle of Calot. A hook cautery is used to carefully incise the peritoneum overlying the triangle of Calot, continuing along the medial aspect of the proximal gallbladder. As the infundibulum is retracted superomedially, peritoneum overlying the posterolateral aspect of the triangle of Calot is similarly incised using hook cautery. All remaining connective tissue is dissected out of the triangle of Calot using blunt dissection and hook cautery as needed to fully mobilize the gallbladder infundibulum.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic gallstones
* Gallstones>3cm in diameter
* Fulfilled gallstones
* Acute or chronic cholecystitis
* Acalculous cholecystitis
* Gallbladder polyps >10mm in diameter
* Symptomatic gallbladder polyps
* Gallbladder stones associated with polyps
* Porcelain gallbladder
* Gallstone pancreatitis

Exclusion Criteria:

* Suspicion of gallbladder cancer
* General condition is poor,inability to tolerate gallbladder cancer
* Important organ dysfunction
* Severe abdominal cavity adhesion
* Bleeding disorders,blood coagulation dysfunction
* Acute cholangitis with serious complications(gallbladder empyema,gangrene,perforation)
* Acute cholangitis
* Pregnancy(first or third trimester)
* Abdominal dysfunction or peritonitis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
complication rate | one month
  biliary injury,artery injury etc.

SECONDARY OUTCOMES:
conversion rate | From date of randomization until the date of first documented progression ,assessed up to 12 months
  The frequency of conversion to open surgery.

OTHER OUTCOMES:
hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1 weeks
  The hospitalization time after operation
blood loss | From date of randomization until the date of first documented progression ,assessed up to 12 months
  the total amount of operation bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Fan yi fang, Prof., Principal Investigator — Department of Hepatobiliary Surgery(I),Zhujiang Hospital
Locations (1):
- Department of Hepatobiliary (I),Zhujiang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Dahmane R, Morjane A, Starc A. Anatomy and surgical relevance of Rouviere's sulcus. ScientificWorldJournal. 2013 Nov 6;2013:254287. doi: 10.1155/2013/254287. eCollection 2013. PMID 24319350